CLINICAL TRIAL: NCT04691193
Title: The Effect of STarT Back Screening Tool in Determining Prognosis and Workforce Loss in Patients With Acute-Subacute Low Back Pain and Its Relationship With Kinesiophobia
Brief Title: The Effect of STarT Back Screening Tool
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, nihal tezel, medical doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: DiskapiYBERH2
Record Dates: First submitted 2020-12-23; First posted 2020-12-31 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Low Back Pain
Keywords: sTart back secreening tool; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study and control group: The study group included patients with low back pain for less than 3 months. The control group consists of healthy volunteers.

SUMMARY:
The aim of this study is to examine the effectiveness of StArt Back Tool test in determining prognosis and loss of workforce in patients presenting with low back pain complaints in the acute-subacute period and to examine the relationship between StArt Back Tool test and kinesophobia.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common disorder that affects about 80% of adults at least once in a period of their life. 10% of low back pain becomes chronic and can affect the quality of life negatively and lead to disability. The STarT-Back-Tool was developed to identify people with poor prognosis, such as difficulty returning to work, loss of work force, disability. It has been reported that it would be beneficial to categorize patients according to their risk levels with this tool and plan treatment in primary care treatment centers. Being able to identify patients with a high probability of becoming chronic in the early period is very important to reduce or prevent disability that may occur. The aim of this study is to examine the effectiveness of StArt Back Tool test in determining prognosis and loss of workforce in patients presenting with low back pain complaints in the acute-subacute period and to examine the relationship between StArt Back Tool test and kinesophobia.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Low back pain for less than 3 months
* Sign the written informed consent.
* Being able to read and write

Exclusion Criteria:

* Inflammatory rheumatologic disease
* Having a history of lumbar surgery
* Back pain for more than 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
STart Back screening Tool | within 6 month
  to measure baseline risk of possible future poor outcome.
Roland Morris Questionnaire | within 6 month
  to determine function

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia | at the beginning
  to determine kinesiophobia

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Tezel, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- DiskapiYBERH, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Forsbrand MH, Grahn B, Hill JC, Petersson IF, Post Sennehed C, Stigmar K. Can the STarT Back Tool predict health-related quality of life and work ability after an acute/subacute episode with back or neck pain? A psychometric validation study in primary care. BMJ Open. 2018 Dec 22;8(12):e021748. doi: 10.1136/bmjopen-2018-021748. PMID 30580256
- [Background] Suri P, Delaney K, Rundell SD, Cherkin DC. Predictive Validity of the STarT Back Tool for Risk of Persistent Disabling Back Pain in a U.S. Primary Care Setting. Arch Phys Med Rehabil. 2018 Aug;99(8):1533-1539.e2. doi: 10.1016/j.apmr.2018.02.016. Epub 2018 Apr 3. PMID 29625095
- [Result] Hill JC, Dunn KM, Lewis M, Mullis R, Main CJ, Foster NE, Hay EM. A primary care back pain screening tool: identifying patient subgroups for initial treatment. Arthritis Rheum. 2008 May 15;59(5):632-41. doi: 10.1002/art.23563. PMID 18438893